CLINICAL TRIAL: NCT03893786
Title: Upper Limb Rehabilitation Using Armeo Spring in Patients With Parkinson's Disease.
Brief Title: Robotic Rehabilitation of Upper Limb in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Professor, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29/2018
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Treatment (Experimental): Fifteen patients with Parkinson's Disease will perform ten 45-minutes training sessions of the upper limb using the Armeo®Spring applied bilaterally, an electromedical device aimed at improving force and coordination in neurologically affected patients.
  The device was built to sustain the forearm during the upper limb training and it is equipped with a VR screen with which the patient may interact during the playful and motivating rehab.
  Interventions: Device: Robotic Rehabilitation
- Conventional Treatment (Active Comparator): Fifteen patients with Parkinson's Disease will undergo ten 45-minutes training sessions of the upper limb with a traditional approach, performing the same excercises of the experimental group, i.e. flexo-extension of the wrist, prono-supination of the forearm, etcc.
  Interventions: Device: Robotic Rehabilitation

INTERVENTIONS:
Device: Robotic Rehabilitation — Fifteen patients with Parkinson's Disease will perform ten 45-minute training sessions of the upper limb bilaterally with the Armeo®Spring, an electromedicad device aimed at improving force and coordination in neurologically affected patients.
  The device was built to sustain the forearm during the upperlimb training and is equipped with a VR screen with which the patient may interact during the playful and motivating rehab.

SUMMARY:
It has been shown that robot-assisted therapy may be considered an effective and reliable method for the delivery of highly repetitive training useful to boost neuroplasticity. Thus, an early, intensive, repetitive and task oriented training could be an ideal strategy to facilitate relearning of motor function and to improve motor function. The ARMEO-S® is a specific upper limb electromedical device mainly used to reduce spasticity and improve muscle force. To date robotic upper limb training has been applied only in patiebts with brain injury and spinal cord lesions.

Aim of the study is to evaluate the efficacy of ARMEO-S in improving upper limb agility in a sample of PD patients, as compared to traditional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD diagnosed according to the UK BRAIN BANK criteria
* Hoehn-Yahr stage 2- 3
* MMSE score ≥ 23

Exclusion Criteria:

* Severe Dyskinesia

  * On-Off Motor fluctuations
  * History of stereotaxic brain surgery for PD;
  * Changes in dopamine therapy dose in any time within 3 months prior to baseline;
  * Any other medical that may compromise the patient's participation in this study such as history of ostheoarthritis or neuropathies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
UPDRS rating scale- Section III | 2 months
  To assess whether PD patients may got better results in the motor part of the UPDRS after the UL training
Nine hole peg test | 2 months
  To evaluate if the patients will get better dexterity after the robotic training

SECONDARY OUTCOMES:
Upper Limb Fugl-Mayer | 2 months
  to verify whether PD patients may present with an increase in muscle strenght after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neurolesi, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: Undecided